CLINICAL TRIAL: NCT06493331
Title: The Effect of the Talking Circle for Pediatric Nursing Students (TC4PN) Activity on Therapeutic Communication Skills
Brief Title: Talking Circle for Pediatric Nursing Students (TC4PN) Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Özge Karakaya Suzan, Principal Investigator, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Talking Circle
Record Dates: First submitted 2024-06-12; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Therapeutic Alliance; Nursing Caries
Keywords: herapeutic communication skills; nurse student; nurse education

STUDY DESIGN:
Who Masked: Participant
Masking Description: participants do not know which group they are in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A workflow diagram will be created according to the gaps in the students' lesson plan, and the groups will create conversation circles and share communication under the leadership of two faculty members (Ö.K.S and E.C). The talking circle application will consist of four sessions. Each talking circle will last 90-120 minutes. At the end of the semester, the 'Therapeutic Communication Skills Scale for Nursing Students' will be administered to the students as a final test.
  Interventions: Other: Talking Circle
- Control (No Intervention): No activity will be applied to control group students during the case collection process. At the end of the semester, the 'Therapeutic Communication Skills Scale for Nursing Students' will be administered as a final test to the students.

INTERVENTIONS:
Other: Talking Circle — step 1 A round seating area is created with chairs. Questions addressing students' perspectives on therapeutic communication styles, the difficulties and conveniences in their communication, and the problems they experience.
  step 2 An object that indicates the talking order will be determined (ball). This object will pass from hand to hand and determine the order of speaking.
  A conversation is started and the students are asked about their thoughts and experiences regarding communication with the pediatric patient and their family with questions prepared by the researchers.
  step 3 The student who does not want to talk can say 1 pass. In the next round, he is encouraged to speak.
  When the sharing is completed, the experiences of the participants will be shared and group comments will be received.
  Arms: Intervention

SUMMARY:
Nursing students communicate with patients during clinical practice to assess their needs and environmental factors affecting their health. However, nursing students often find therapeutic communication to be one of the most stressful tasks. Specifically, studies report that nursing students face difficulties in communicating to care for pediatric patients.

In this regard, the aim of this research is; To examine the effects of Talking Circle activities based on JOHN LOWE's self-confidence theory on the therapeutic communication skills of pediatric nursing students.

DETAILED DESCRIPTION:
Nursing students communicate with patients during clinical practice to assess their needs and environmental factors affecting their health. However, nursing students often find therapeutic communication to be one of the most stressful tasks. In particular, studies report that nursing students face difficulties in communicating to care for pediatric patients. Communication is situational and contextual and can be influenced by factors such as patient characteristics.

Therapeutic communication is an intentional interaction aimed at improving the emotional and physical well-being of the patient. This communication is associated with the success of professions that focus on supporting people. Nursing is a profession that spends most of its professional life providing patient care. Effective therapeutic communication is essential for optimal nursing practice regardless of employment setting. Therapeutic communication aims to create quality health care based on awareness, empathy and trust between the nurse and the patient. Research shows that effective communication between patients and nurses increases patient satisfaction and quality of care and reduces the length of hospital stay. It is reported that inadequate or negative communication poses health risks for the patient.

Healthcare professionals report that communicating with hospitalized children is challenging. In this context, it is important to teach students how to communicate effectively with children and family members in the Child Health and Diseases Nursing Course, which teaches care and communication to children. Current literature emphasizes that the curriculum should be expanded with practices that will improve the effective communication skills of nursing students.

Although it is stated that therapeutic communication is necessary for effective child-centered care in all healthcare settings, the training provided to nurses on encouraging and strengthening nurse-child communication is unfortunately inadequate. Nursing education aims to train nurses with strong communication skills.Therefore, in nursing education, nursing students need to discover strategies that will enable them to understand therapeutic communication in depth and acquire skills that will enable them to communicate effectively with patients after graduation.

In this regard, the aim of this research is; To examine the effects of Talking Circle activities based on JOHN LOWE's self-confidence theory on the therapeutic communication skills of pediatric nursing students.

ELIGIBILITY:
Inclusion Criteria:

* Third-year nursing students must fill out the data collection tools,
* Take the Effective Communication and Human Behavior course in their first year,
* Pass all semester courses successfully,
* Volunteer to participate in the research.

Exclusion Criteria:

* Failure to complete data collection tools
* Withdrawing from the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-04-26 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Therapeutic Communication Skills Scale | Baseline, (1st measurement) -immediately after the intervention (2nd measurement)
  Between-group differences in Therapeutic Communication Skills Scale for Nursing Students scores
  Therapeutic Communication Skills Scale for Nursing Students
  The scale consists of 16 items and 3 sub-dimensions: "Non-therapeutic Communication Skills", "Therapeutic Communication Skills-1", "Therapeutic Communication Skills-2". The first sub-dimension of the scale consists of 7 items, the second sub-dimension consists of 6 items, and the third sub-dimension consists of 3 items. The scale is a 7-point Likert type ranging from 1 to 7, and there are no reverse coded items in the scale. The highest score that can be obtained from the scale is 16x7=112, and the lowest score is 16x1=16. The increase in scale scores shows that communication skills have increased.

CONTACTS AND LOCATIONS:
Overall Officials: Nursan ÇINAR, PhD, Principal Investigator — SAKARYA UNİVERSITY; Emine Cincioglu, PhD, Principal Investigator — Sakarya University
Locations (1):
- sakarya University, Sakarya, Serdivan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
AFTER THE ARTICLE IS ACCEPTED IN A JOURNAL, IT MAY BE PUBLICLY AVAILABLE.